CLINICAL TRIAL: NCT01292083
Title: A Pilot Clinical Trial to Evaluate the Biological Activity of 5-azacitidine on ER and PR Expression in Triple Negative Invasive Breast Cancer
Brief Title: Azacitidine in Treating Patients With Triple Negative Stage I-IV Invasive Breast Cancer That Can Be Removed By Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No accrual last 2 years
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1B-09-15; NCI-2011-00117 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-02-02; First posted 2011-02-09 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Recurrent Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer; Triple-negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Azacitidine; Immunohistochemistry; Polymerase Chain Reaction; Blotting, Western; Base Sequence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): See Detailed Description
  Interventions: Drug: azacitidine; Other: laboratory biomarker analysis; Other: immunohistochemistry staining method; Genetic: polymerase chain reaction; Genetic: western blotting; Genetic: nucleic acid sequencing; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: azacitidine — Given IV
  Other Names: 5-AC; 5-azacytidine; azacytidine; Vidaza
Other: laboratory biomarker analysis — Correlative studies
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Genetic: polymerase chain reaction — Correlative studies
  Other Names: PCR
Genetic: western blotting — Correlative studies
  Other Names: Blotting, Western; Western Blot
Genetic: nucleic acid sequencing — Correlative studies
  Other Names: Gene Sequencing; Molecular Biology, Nucleic Acid Sequencing
Procedure: therapeutic conventional surgery — Undergo definitive breast surgery

SUMMARY:
This clinical trial studies azacitidine in treating patients with triple negative stage I-IV invasive breast cancer that can be removed by surgery. Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To evaluate the ability of deoxyribonucleic acid (DNA) methylation inhibition using 5-azacitidine to induce expression of the estrogen receptor (ER) and progesterone receptor (PR) genes in solid human triple negative invasive breast cancer. SECONDARY OBJECTIVES: I. To determine the effect of systemic 5-azacitidine therapy on the expression of other methylated genes in triple negative invasive breast cancer using an Illumina GoldenGate array. OUTLINE: Patients receive azacitidine intravenously (IV) over 10-40 minutes 5 days a week for 2 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo definitive breast surgery within 12 days of the last dose of azacitidine.

ELIGIBILITY:
Inclusion Criteria:

* Resectable tumor measuring 2 cm or more
* Histologically documented triple negative invasive breast cancer characterized by 0% Immunohistochemistry (IHC) nuclear staining for ER-alpha, 0% IHC nuclear staining for PR-alpha, and no amplification of HER2/neu by fluorescence in situ hybridization (FISH); standard IHC assays for ER and PR use antibodies to ER-alpha and PR-alpha and PR-beta
* Southwest Oncology Group (SWOG) performance status of less than or equal to 1
* Absolute neutrophil count (ANC) >= 1500/μL
* Hemoglobin (Hgb) >= 9 g/dL
* Platelets >= 100,000/uL
* Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamic pyruvate transaminase (SGPT) =< 2.5 x upper limit normal (ULN) or =< 5.0 x ULN in patients with liver metastases
* Creatinine =< 2.0 mg/dL Or Calculated Creatinine Clearance >= 50 ml/min
* Albumin >= 3 g/dL
* Potassium >= lower limit normal (LLN)
* Phosphorous >= LLN
* Calcium >= LLN
* Magnesium > LLN
* Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to start of treatment
* Accessible for treatment and follow-up
* Written informed consent prior to study entry

Exclusion Criteria:

* HER2/neu amplification by FISH
* Concurrent neoadjuvant treatment with chemotherapy, endocrine therapy, or radiotherapy
* Known hypersensitivity to azacitidine or mannitol
* Preexisting hepatic impairment or renal impairment
* Intent to receive additional neoadjuvant therapy prior to surgery
* Concurrent use of an histone deacetylase (HDAC) inhibitor or hydralazine
* Known diagnosis of human immunodeficiency virus (HIV) infection
* Major surgery < 4 weeks prior to starting study drug
* Pregnant or breastfeeding or female of reproductive potential not using an effective method of birth control
* Other concurrent severe, uncontrolled infection or intercurrent illness, including but not limited to ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements
* Prior antiestrogens (selective estrogen receptor modulator [SERM] or aromatase inhibitors) within 6 months of study entry
* Underlying medical, psychiatric or social conditions that would preclude patient from receiving treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Percent of participants with ER/PR response after receiving 10 doses of 5-Azacitidine | 6 months after enrollment of last patient

CONTACTS AND LOCATIONS:
Overall Officials: Agustin Garcia, MD, Principal Investigator — University of Southern California